CLINICAL TRIAL: NCT03239483
Title: A Randomized, Double Blind, Placebo-Controlled, Phase 1 Safety and Pharmacokinetic Study of Dapivirine Gel (0.05%) Administered Rectally to HIV-1 Seronegative Adults
Brief Title: Safety and Pharmacokinetic Study of Dapivirine Gel (0.05%) Administered Rectally to HIV-1 Seronegative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTN-026; 12021 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Results first posted 2019-11-07 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2019-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapivirine gel (Experimental): Participants will receive a single dose of dapivirine gel rectally, followed by 7 daily doses of dapivirine gel to be administered under direct observation in the clinic.
  Interventions: Drug: Dapivirine gel
- Placebo gel (Placebo Comparator): Participants will receive a single dose of placebo gel rectally, followed by 7 daily doses of placebo gel to be administered under direct observation in the clinic.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Dapivirine gel — Dapivirine gel (0.05%); administered rectally
  Arms: Dapivirine gel
Drug: Placebo gel — Universal HEC placebo gel; administered rectally
  Arms: Placebo gel

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics (PK) of dapivirine gel (0.05%) administered rectally to HIV-1 seronegative adults.

DETAILED DESCRIPTION:
This study will evaluate the safety and pharmacokinetics (PK) of dapivirine gel (0.05%) administered rectally to HIV-1 seronegative adults.

Participants will be randomized to receive a single dose of either rectally administered dapivirine gel (0.05%) or placebo gel at study entry (Day 0). Following a minimum 2-week washout period, participants or study staff will administer daily rectal doses of the assigned gel for 7 consecutive days under direct observation in the clinic.

Participants will be in the study for approximately 40 days, and they will attend 16 study visits. Study visits may include behavioral assessments, physical examinations, blood and urine collection, and pelvic and anorectal sample collection. Some visits will include intensive PK sampling. Study staff will contact participants 1 week after Visit 16 for follow-up safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 45 years (inclusive) at Screening, verified per site standard operating procedure (SOP)
* Able and willing to provide written informed consent
* HIV-1/2 uninfected at Screening and Enrollment, per applicable algorithm in Appendix II of the protocol and willing to receive HIV test results
* Able and willing to provide adequate locator information, as defined in site SOP
* Available to return for all study visits and willing to comply with study participation requirements
* In general good health at Screening and Enrollment, as determined by the site Investigator of Record (IoR) or designee
* Per participant report, a history of consensual receptive anal intercourse (RAI) at least once in the past calendar year
* Willing to not take part in other research studies involving drugs, medical devices, genital or rectal products, or vaccines for the duration of study participation, including the time between Screening and Enrollment
* Willing to be sexually abstinent for 72 hours prior to each study visit, during the study product use periods and for 72 hours after biopsy collection. Note: See Criteria 12 and 13 for additional restrictions for female participants
* Willing to abstain from inserting any non-study products into the rectum for 72 hours prior to each study visit and during the study product use periods. Note: See Criteria 12 and 13 for additional restrictions for female participants

Females must also meet the following additional inclusion criteria to be eligible for study inclusion:

* Women over the age of 21 (inclusive) must have documentation of a satisfactory Pap within the past 3 years prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result
* Willing to be sexually abstinent for 72 hours prior to each study visit and during the study product use periods and for 7 days after biopsy collection
* Willing to abstain from inserting any non-study products into the vagina for 72 hours prior to each study visit, during the study product use periods and for 7 days after biopsy collection
* Willing to use an effective method of contraception for at least 30 days (inclusive) prior to Enrollment and intending to continue use of an effective method for the duration of study participation; effective methods include: hormonal methods (except contraceptive ring), intrauterine device (IUD), sterilization (of participant and/or partner, as defined in site SOPs), or sexually abstinent for 90 days prior to Screening

Exclusion Criteria:

* At Screening:

  * Hemoglobin Grade 1 or higher*
  * Platelet count Grade 1 or higher*
  * White blood count Grade 2 or higher*
  * Serum creatinine greater than 1.3× the site laboratory upper limit of normal (ULN)
  * International normalized ratio (INR) greater than 1.5× the site laboratory ULN
  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher*
  * Positive for hepatitis C antibody
  * Positive for hepatitis B surface antigen
  * History of inflammatory bowel disease by participant report
  * *As per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017
  * Note: Otherwise eligible participants with an exclusionary test result (other than HIV, HBV or HCV) can be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
* Anticipated use of and/or unwillingness to abstain from the following medications during study participation:

  * Heparin, including Lovenox®
  * Warfarin
  * Plavix® (clopidogrel bisulfate)
  * Aspirin (greater than 81 mg)
  * Non-steroidal anti-inflammatory drugs (NSAIDS)
  * Any other drugs that are associated with increased likelihood of bleeding
  * CYP3A inducer(s) and/or inhibitor(s) as specified in the MTN-026 Study-Specific Procedures (SSP) Manual
  * Hormone-replacement therapy in tablet, injectable or gel form
* Known adverse reaction to any of the components of the study products
* Use of post-exposure prophylaxis (PEP) for potential HIV exposure within the 6 months prior to Enrollment
* Use of pre-exposure prophylaxis (PrEP) for HIV prevention within the 6 months prior to Enrollment, and/or anticipated use during trial participation
* Use of systemic immunomodulatory medications within the 6 months prior to Enrollment, and/or anticipated use during trial participation
* RAI without a condom and/or penile-vaginal intercourse with a partner who is known to be HIV-positive in the past 6 months
* Non-therapeutic injection drug use in the 12 months prior to Screening and Enrollment
* Participation in research studies involving drugs, medical devices, genital or rectal products, or vaccines within 45 days of the Enrollment Visit
* At Screening, participant report of treatment for an anogenital STI within the past 3 months
* At Screening, participant-reported symptoms and/or clinical or laboratory diagnosis of active anorectal or reproductive tract infection requiring treatment per current World Health Organization (WHO) guidelines (http://www.who.int/hiv/pub/sti/pub6/en/) or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic Neisseria gonorrhea (GC), Chlamydia trachomatis (CT) infection, syphilis, active herpes simplex virus (HSV) lesions, anogenital sores or ulcers, or symptomatic genital warts, cervicitis, chancroid, pelvic inflammatory disease (PID), bacterial vaginosis (BV), symptomatic vaginal candidiasis, other vaginitis, trichomoniasis. Note: Otherwise eligible participants with an exclusionary UTI, BV and/or candida finding may be re-tested during the screening process.
* At Enrollment, active anorectal or reproductive tract infection requiring treatment per current WHO guidelines (http://www.who.int/hiv/pub/sti/pub6/en/) or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic GC, CT, syphilis, active HSV lesions, anogenital sores or ulcers, symptomatic genital warts, bacterial vaginosis, symptomatic vaginal candidiasis, other vaginitis, trichomoniasis, chancroid, cervicitis and PID. Note: HSV-1 or HSV-2 seropositive diagnosis with no active lesions is permitted since treatment is not required
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Females who meet any of the following additional criteria will be excluded from the study:

* Pregnant or breastfeeding at either Screening or Enrollment or intends to become pregnant or start breastfeeding during study participation. Note: A documented negative pregnancy test performed by study staff is required for inclusion; however, a self-reported pregnancy is adequate for exclusion from screening/enrollment into the study.
* Last pregnancy outcome 90 days or less prior to Screening
* Has had a hysterectomy
* At Enrollment, has a clinically apparent Grade 1 or higher pelvic exam finding (observed by study clinician or designee) per the Female Genital Grading Table for Use in Microbicide Studies [Addendum 1, Dated November 2007]. Note: Cervical friability bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross D. Cranston, MD, FRCP, Study Chair — Fundació Lluita Contra la Sida, Hospital Universitari Germans Trias I Pujol
Locations (3):
- United States (2):
  - Alabama CRS, Birmingham, Alabama
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
- Silom Community Clinic CRS, Nonthaburi, Bangkok, Thailand

REFERENCES:
- [Derived] Bauermeister JA, Tingler RC, Dominguez C, Dunne EF, Hoesley C, Ho K, Johnson S, Lucas J, Macagna N, Brown E, Gundacker H, Peda M, Jacobson CE, Kramzer L, Singh D, Dezzutti CS, Ayudhya RPKN, Marzinke MA, Piper J, Devlin B, Nuttall J, McGowan I, Hendrix CW, Cranston RD; MTN 026 team. Acceptability of a Dapivirine/Placebo Gel Administered Rectally to HIV-1 Seronegative Adults (MTN-026). AIDS Behav. 2022 May;26(5):1333-1346. doi: 10.1007/s10461-021-03490-8. Epub 2021 Oct 17. PMID 34657218
- [Derived] Cranston RD, Brown E, Bauermeister J, Dunne EF, Hoesley C, Ho K, Johnson S, Lucas J, Dominguez-Islas C, Gundacker H, Peda M, Jacobson CE, Kramzer L, Singh D, Dezzutti CS, Kunjara Na Ayudhya RP, Brand RM, Wang L, Marzinke MA, Piper J, Devlin B, Nuttall J, McGowan I, Hendrix CW. A Randomized, Double Blind, Placebo-Controlled, Phase 1 Safety, and Pharmacokinetic Study of Dapivirine Gel (0.05%) Administered Rectally to HIV-1 Seronegative Adults (MTN-026). AIDS Res Hum Retroviruses. 2022 Apr;38(4):257-268. doi: 10.1089/AID.2021.0071. Epub 2021 Dec 6. PMID 34498980

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapivirine Gel | Placebo Gel
Started (one participant withdrew consent and did not receive any study product) | 19 | 9
Completed | 17 | 9
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapivirine Gel | Placebo Gel | Total
Number analyzed (Participants) | 19 | 9 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 9 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 26 [18 to 42] | 35 [21 to 40] | 33 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 15 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 11 | 2 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19
  Thailand | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Grade 2 or Higher Adverse Events (AEs)
Description: As defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 1, 2 and 3 (Female Genital [Dated November 2007], Male Genital [Dated November 2007] and Rectal [Clarification Dated May 2012] Grading Tables for Use in Microbicide Studies)
Time Frame: Measured after the participant has started study product until the participant's study termination at approximately Day 40
Population: enrolled participants receiving at least one dose of study product
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Gel | Placebo Gel
Number analyzed (Participants) | 18 | 9
Participants | 3 | 5
Statistical Analysis 1: Comparison: Dapivirine Gel vs Placebo Gel; two-sided Fisher's Exact Test; Test type: Superiority; p = 0.072, Fisher Exact

2. Primary Outcome: Measurement of Dapivirine Concentrations in Plasma
Description: As assessed by pharmacokinetic sampling and analysis
Time Frame: Sample collected at approximately 1, 2, 24, 48 and 72 hours after first single dose, 24 hours after first dose during daily dosing, before last dose and 1,2, 24,48, and 72 hours after last dose.
Population: enrolled participants on the Dapivirine arm who received at least one dose of study product and had a sample collected at the specific time-point. 0 is an estimate for values below the limit of quantification (LLOQ = 20 pg/mL) since only numeric values are allowed. The value would be somewhere between the LLOQ and 0.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Dapivirine Gel
Number analyzed (Participants) | 18
pg/mL
  30 to 60 minutes after single dose | 31.5 [0 to 54.6]
  120 minutes after single dose: number analyzed (Participants) | 10
  120 minutes after single dose | 326 [153 to 481]
  24 hours after single dose | 20.1 [0 to 56.6]
  48 hours after single dose | 0 [0 to 27.3]
  72 hours after single dose | 0 [0 to 0]
  24 hours after first daily dose | 67.9 [43.1 to 111.0]
  Before last daily dose: number analyzed (Participants) | 17
  Before last daily dose | 167 [136 to 219]
  30 to 60 minutes after last daily dose: number analyzed (Participants) | 8
  30 to 60 minutes after last daily dose | 290.5 [147.0 to 506.5]
  120 minutes after last daily dose: number analyzed (Participants) | 9
  120 minutes after last daily dose | 403 [330 to 493]
  24 hours after last daily dose: number analyzed (Participants) | 17
  24 hours after last daily dose | 119.0 [86.4 to 172.0]
  48 hours after last daily dose: number analyzed (Participants) | 17
  48 hours after last daily dose | 113 [69 to 132]
  72 hours after last daily dose: number analyzed (Participants) | 17
  72 hours after last daily dose | 80.3 [47.3 to 129.0]

3. Primary Outcome: Measurement of Dapivirine Concentrations in Rectal Fluid
Description: As assessed by pharmacokinetic rectal fluid sampling and analysis
Time Frame: Sample collected at approximately 1, 2, 24, 48 and 72 hours after first single dose, 24 hours after first dose during daily dosing, and 1,2, 24,48, and 72 hours after last dose.
Population: enrolled participants on the Dapivirine arm who received at least one dose of product and had a sample collected at the specific time-point. 0 is an estimate for values below the limit of quantification (LLOQ = 0.001 ng/mg) since only numeric values are allowed. The value would be somewhere between the lower limit of quantification and 0.
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | Dapivirine Gel
Number analyzed (Participants) | 18
ng/mg
  30 to 60 minutes after first application: number analyzed (Participants) | 8
  30 to 60 minutes after first application | 30.1 [16.1 to 43.9]
  120 minutes after single dose: number analyzed (Participants) | 8
  120 minutes after single dose | 12.765 [6.055 to 141.500]
  24 hours after single dose: number analyzed (Participants) | 8
  24 hours after single dose | 0 [0 to 0.016]
  48 hours after single dose: number analyzed (Participants) | 4
  48 hours after single dose | 0.009 [0 to 0.038]
  72 hours after single dose: number analyzed (Participants) | 6
  72 hours after single dose | 0 [0 to 0]
  24 hours after first daily dose | 0.180 [0 to 1.910]
  30 to 60 minutes after last daily dose: number analyzed (Participants) | 7
  30 to 60 minutes after last daily dose | 89.7 [44.9 to 258.0]
  120 minutes after last daily dose: number analyzed (Participants) | 8
  120 minutes after last daily dose | 26.65 [4.95 to 278.50]
  24 hours after last daily dose: number analyzed (Participants) | 7
  24 hours after last daily dose | 0.007 [0 to 0.096]
  48 hours after last daily dose: number analyzed (Participants) | 4
  48 hours after last daily dose | 0 [0 to 0.042]
  72 hours after last daily dose: number analyzed (Participants) | 6
  72 hours after last daily dose | 0 [0 to 0.013]

4. Primary Outcome: Measurement of Dapivirine Concentrations in Rectal Mucosal Tissue Homogenates
Description: As assessed by pharmacokinetic rectal mucosal tissue homogenates sampling and analysis
Time Frame: Sample collected at approximately 1, 2, 24, 48 and 72 hours after first single dose and 1,2, 24,48, and 72 hours after last dose.
Population: enrolled participants on the Dapivirine gel arm who received at least one dose of study product and had a sample collected at the specific time-point. 0 is an estimate for values below the limit of quantification (LLOQ = 0.001 ng/mg) since only numeric values are allowed. The value would be somewhere between the LLOQ and 0.
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | Dapivirine Gel
Number analyzed (Participants) | 18
ng/mg
  30 to 60 minutes after single dose: number analyzed (Participants) | 8
  30 to 60 minutes after single dose | 0.256 [0 to 0.666]
  120 minutes after single dose: number analyzed (Participants) | 10
  120 minutes after single dose | 0 [0 to 0.600]
  24 hours after single dose: number analyzed (Participants) | 8
  24 hours after single dose | 0 [0 to 0]
  48 hours after single dose: number analyzed (Participants) | 4
  48 hours after single dose | 0 [0 to 0]
  72 hours after single dose: number analyzed (Participants) | 6
  72 hours after single dose | 0 [0 to 0]
  30 to 60 minutes after last daily dose: number analyzed (Participants) | 7
  30 to 60 minutes after last daily dose | 0 [0 to 0]
  120 minutes after last daily dose: number analyzed (Participants) | 8
  120 minutes after last daily dose | 0 [0 to 0.151]
  24 hours after last daily dose: number analyzed (Participants) | 7
  24 hours after last daily dose | 0 [0 to 0]
  48 hours after last daily dose: number analyzed (Participants) | 3
  48 hours after last daily dose | 0 [0 to 0]
  72 hours after last daily dose: number analyzed (Participants) | 6
  72 hours after last daily dose | 0 [0 to 0]

5. Primary Outcome: Terminal Half-life of Dapivirine Concentrations in Plasma
Description: The terminal half-life of dapivirine in plasma samples was estimated by fitting a linear regression on the log-transformed concentrations from the 24, 48 and 72 hour time-points after the single and multiple doses.Each regression model includes an adjustment for the difference in concentration after multiple dosing. For each participant, Beta was calculated as the negative of the slope of their repression and half-life was log(2)/Beta. Due to the large number of concentrations below the limit of quantification after the single dose, the estimateion of Beta and half-life relied only on concentration after the multiple dosing for most of the participants.
Time Frame: From samples collected 24 hours after first dose to 72 hours after last daily dose
Population: enrolled participants on the Dapivirine gel arm who received at least one dose of study product. One participant with a negative estimate for the elimination rate due to an increasing trend in their concentration after multiple dosing and one participant with no values above the limit of quantification were excluded.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dapivirine Gel
Number analyzed (Participants) | 16
hours | 52.6 [35.3 to 86.2]

6. Secondary Outcome: Acceptability: Ease of Use
Description: The number of participants who responded by questionnaire that the study product was easy or very easy to use.
Time Frame: after completing the study (study day 40)
Population: All enrolled participants who completed the exit behavioral questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Gel | Placebo Gel
Number analyzed (Participants) | 17 | 9
Participants | 16 | 9
Statistical Analysis 1: Comparison: Dapivirine Gel vs Placebo Gel; Test type: Superiority; p = 1.00, Fisher Exact — This is a calculated p-value. P-values of 1.0 are possible when using the Fisher Exact test method

7. Secondary Outcome: Acceptability: Comfort
Description: The number of participants who responded on a questionnaire that the study product was comfortable or very comfortable.
Time Frame: after completing the study (study day 40)
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Gel | Placebo Gel
Number analyzed (Participants) | 17 | 9
Participants | 15 | 7
Statistical Analysis 1: Comparison: Dapivirine Gel vs Placebo Gel; Test type: Superiority; p = 0.591, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion (between 40 to 86 days).
Arm/Group | Dapivirine Gel | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/9
Other Adverse Events (participants affected / at risk) | 6/18 | 7/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Gel (N=18) | Placebo Gel (N=9)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
blood pressure increased (Investigations) | 1 (2) | 0 (0)
coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03239483/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03239483/SAP_001.pdf